CLINICAL TRIAL: NCT00658840
Title: A Phase II Study of Concurrent Chemo-radiotherapy With Capecitabine for Unresectable Locally Advanced Pancreatic Carcinoma
Brief Title: Concurrent Chemo-radiotherapy With Capecitabine for Unresectable Locally Advanced Pancreatic Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Tae Hyun Kim, National Cancer Center Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-199
Record Dates: First submitted 2008-03-24; First posted 2008-04-15 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Immobilization

ARMS (1):
- 1 (Experimental): Primary objectives :
  To evaluate the tumor response rate, local control rate and compliance (acute and late toxicity, esp. gastrointestinal tract toxicity) of concurrent chemo-radiotherapy with oral capecitabine in patients with unresectable locally advanced pancreatic carcinoma
  Secondary objectives :
  To evaluate the impact of concurrent chemo-radiotherapy with oral capecitabine in patients with unresectable locally advanced pancreatic carcinoma by analyzing the progression-free survival rate and overall survival rate.
  Interventions: Drug: Capecitabine (Xeloda®); Radiation: Localization, simulation and immobilization

INTERVENTIONS:
Drug: Capecitabine (Xeloda®) — Capecitabine is administered orally at a dose of 800 mg/m2 twice daily (total daily dose 1600mg/ m2) continuous regimen regimen during RT (5 days of treatment followed by a 2 day rest: Saturday and Sunday). Capecitabine is given approximately 12 hours apart and taken orally with water within 30 minutes after ingestion of food (breakfast or dinner).
Radiation: Localization, simulation and immobilization — Radiation dose and planning
  1. Total dose 55.8Gy, 28 fractions, 6-7 weeks (1.8 Gy/day). A cone down after 45 Gy will be performed to emcompass GTV with a margin of 1-1.5cm.
  2. Dose prescription : 90% isodose volume of prescribed dose encompassed PTV
  3. The dose-volume histogram (DVH) of targets, such as GTV, CTV, and PTV, and the normal tissues, such as the liver, duodenum, stomach, the kidneys, spinal cord, etc., was calculated.

SUMMARY:
The only curative option for pancreatic cancer patients is surgery, but the patients within 20% of them are possible for a radical surgery. Accordingly, concurrent chemo-radiation therapy is generally used for palliation of unresectable pancreatic cancer patients. So far, the use of 5-fluorouracil (5-FU) was the traditional method of chemotherapy. However, these days, oral anti-cancer medicine, capecitabine(Xeloda®), was developed and considered as an alternative medicine of 5-fluorouracil (5-FU). Furthermore, according to the recent results of clinical trials, the clinical use of capecitabine(Xeloda®) with radiation therapy was proved to be very effective and safe. The purpose of this trial is to improve the therapeutic effects by using proton therapy and chemotherapy concurrently.

ELIGIBILITY:
Inclusion Criteria:

* There is no evidence of metastatic disease in the major viscera and no peritoneal seeding
* Patients with biliary or gastroduodenal obstruction must have drainage prior to starting chemoradiation
* All malignant disease must be encompassable within a single irradiation field (15x15cm maximum)
* All patients must have radiographically assessable disease
* No previous irradiation to the planned field
* Age of ≥18 years
* performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score
* Required Entry Laboratory Parameters WBC count ≥ 2,000/mm3;(ANC>1,000), hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 100,000/mm3; total bilirubin ≤ 3.0 mg/dL (Patients with elevated bilirubin due to obstruction should be stented and their bilirubin should be decreas ≤ 3.0 mg/dL prior to study entry); creatinine ≤ 3.0 mg/dL
* Oral intake (including J-tube feeding) of ≥ 1,500 calories/day should be maintained.

Exclusion Criteria:

* There is evidence of metastasis in the major viscera or peritoneal seeding.
* Age of <18 years
* Previous history of RT adjacent to planned field
* poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* pregnant or breast feeding status
* previous history of uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2006-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | two year

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea